CLINICAL TRIAL: NCT04118075
Title: Post Transplantation Cyclophosphamide With or Without Low-dose ATG for Patients With Lymphoid Malignancies Undergoing Allogeneic Stem Cell Transplantation
Brief Title: PT-CY With or Without Low-dose ATG for Lymphoid Malignancies Undergoing Allo-HSCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiong HU, Head, Blood & Marrow Transplantation Program, Chief physician, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RJH-Lym-2018
Record Dates: First submitted 2019-10-04; First posted 2019-10-08 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: GVHD, Acute
Keywords: aGVHD, cGVHD, PT-CY
MeSH Terms: conditions — Graft vs Host Disease; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PT-CY-FK +/- ATG (Experimental): GVHD prophylaxis: PT-CY followed by tacrolimus for all patients. low-dose ATG for patients with unrelated or haplo-identical transplantation.
  Interventions: Drug: PT-CY-FK +/-ATG

INTERVENTIONS:
Drug: PT-CY-FK +/-ATG — GVHD prophylaxis: PT-CY followed by tacrolimus for all patients. low-dose ATG for patients with unrelated or haplo-identical transplantation.
  Other Names: RJH-Lym-2018

SUMMARY:
All patients received Flu-BU-VP16 as myeloablative conditioning followed by cyclophosphamide (D+3 and +4) and subsequent tacrolimus. For patients with unrelated or haplo-donor received low-dose ATG at Day +15.

DETAILED DESCRIPTION:
For patients with high-risk lymphoid malignancies, patients will undergo allo-HSCT from HLA matched sibling, unrelated (9~10/10) donor or hallo-identical donors. For all patients will receive myeloablative conditioning with 5-day fludarabine, 2-day VP-16 and 3-day busulifan. For prophylaxis graft versus host disease (GVHD), patients will receive cyclophosphamide 50mg/kg daily on D+3 and +4 with subsequent tacrolimus starting at D+5. For patients receiving HSCT from unrelated or haplo-donor, low-dose ATG 2.5mg/kg will be given on Day +15.

ELIGIBILITY:
Inclusion Criteria:

* patients with lymphoid malignancies: CR1 or CR2 for acute lymphoblastic leukemia; T cell lymphoma (any CR/PR); B cell lymphoma (PR1 or CR2), hodgkin's disease (CR2 or beyond), Sezary syndrome
* patients with HLA matched sibling, unrelated (HLA 9~10/10 matched) or haplo-identical donor

Exclusion Criteria:

* patients with active infection
* patients with abnormal liver function damage: ALT/AST above 2X normal range
* patients with abnormal renal function damage Scr>160µmol/L;
* patients with insufficient pulmonary function (FEV1，FVC，DLCO<50%）and heart failure or with EF <50%)
* patients with mental instability
* unwilling to give inform consent

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
grade II-IV acute GVHD | Day 100
  cumulated incidence of grade II-IV aGVHD

SECONDARY OUTCOMES:
grade III-IV acute GVHD | Day 100
  cumulated incidence of grade III-IV aGVHD
Non relapse mortality (NRM) | Day 100
  cumulated incidence of NRM
chronic GVHD (cGVHD) | 1 year
  cumulated incidence of overall cGVHD
moderate to sever chronic GVHD | 1 year
  cumulated incidence of moderate to severe cGVHD
relapse rate | 1 year
  cumulated incidence of bone marrow or PET/biopsy documented relapse
non relapse mortality | 1 year
  cumulated incidence of NRM
overall survival | 1 year
  overall survival from entry of study to any cause of death
GVHD-free relapse free survival (GRFS) | 1 year
  survival without II-IV aGVHD, moderate to severe cGVHD, relapse or any other death event of any case

CONTACTS AND LOCATIONS:
Overall Officials: Jiong Hu, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Rui Jin Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Jiang JL, Gao WH, Wang LN, Wan M, Wang L, Hu J. Post-transplantation Cyclophosphamide, Tacrolimus and Low-Dose ATG as GVHD Prophylaxis for Allogeneic Peripheral Stem Cell Transplantation for Adult Patients With Lymphoid Malignancies: A Single Arm Phase II Study. Front Med (Lausanne). 2021 Mar 18;8:630160. doi: 10.3389/fmed.2021.630160. eCollection 2021. PMID 33816524